CLINICAL TRIAL: NCT03670927
Title: Etiosarc: Study of the Environmental Aetiology (Environment, Occupations and Lifestyle) of Sarcomas (Soft Tissue, Visceral and Bone) From a Multicenter French Population-based Case-control Study Among Adults.
Brief Title: Etiosarc: Environmental Aetiology of Sarcomas From a Multicenter French Population-based Case-control Study Among Adults
Acronym: ETIOSARC
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C17-03
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Sarcoma; Environmental Exposure; Occupational Exposure; Life Style
MeSH Terms: conditions — Sarcoma | interventions — Environment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each participant will be asked to provide a salivary sample in order to obtain germline DNA. Salivary samples will be collected by the subjects themselves under instructions from the CRA, using DNA Genotek Oragene 575 collection kit. After collection, samples will be sent at the Biological Resources Center of the Bordeaux hospital university center "Bordeaux Biothèque Santé" for storage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases (incident patients with a diagnosis of primary sarcoma and histologically confirmed by an expert pathologist of the RRePS or ResOs networks in the 15 districts of France participating to this study) Environmental, occupational and lifestyle-related exposures
  Interventions: Other: Environmental, occupational and lifestyle-related exposures
- Controls: Subjects never diagnosed with a primary sarcoma and individually-matched by sex, age (5-years group), and districts of residence and randomly selected from electoral list.
  Environmental, occupational and lifestyle-related exposures
  Interventions: Other: Environmental, occupational and lifestyle-related exposures

INTERVENTIONS:
Other: Environmental, occupational and lifestyle-related exposures — A standardized questionnaire will be administered by a trained interviewer in order to gather information about occupational and residential history, demographic and socioeconomic characteristics and lifestyle factors. At the end of the interview, a saliva sample will be systematically proposed

SUMMARY:
Introduction: Sarcomas are rare tumors of connective tissue. The exact overall incidence of sarcomas is unknown due to diagnostic difficulties and the various histological subtypes (over 80 subtypes). However, the apparent increasing incidence of sarcomas suggests environmental causes such as pesticides. Except for some specific factors (i.e. ionizing radiation, vinyl chloride, dioxin, and genetic predispositions) the scientific knowledge on the aetiology of sarcomas is sparse and inconsistent. France is a particularly appropriate country to set up a study investigating the causes of sarcoma occurrence due to the French organization in treatment and care of sarcoma patients, which is highly structured and revolved around national expert networks. The main objective of the ETIOSARC project is to study the role of lifestyle, environmental and occupational factors in the occurrence of sarcomas among adults from a multicentric population-based case-control study.

Methods and analysis: Cases will be all incident cases (older than 18 years old) identified in 15 districts of France covered by a cancer registry and/or a reference center in sarcoma's patient care over a three-year period with an inclusion start date ranging from the 1st October 2018 to the 1st January 2020 and histologically confirmed by a second review of the diagnosis. Two controls will be individually-matched by sex, age (5-years group), and districts of residence and randomly selected from electoral list. A standardized questionnaire will be administered by a trained interviewer in order to gather information about occupational and residential history, demographic and socioeconomic characteristics and lifestyle factors. At the end of the interview, a saliva sample will be systematically proposed.

This study will permit to validate or not already suspected risk factors for sarcomas such as phenoxyherbicides, chlorophenol and to generate new hypothesis to increase our understanding about the genetic and environmental contributions in the carcinogenicity process.

DETAILED DESCRIPTION:
The main objective of the ETIOSARC study is to assess the role of lifestyle, environmental and occupational factors in the occurrence of sarcomas among adults from a multicenter population-based case-control study.

Specific objectives are:

* To identify environmental risk factors for sarcomas as a whole and for the most frequent subtypes;
* To investigate the interactions between gene polymorphisms and environmental exposures in sarcoma susceptibility;
* To assess whether some specific genetic characteristics of sarcoma' tumors are associated with environmental exposures; We will also explore the feasibility of classifying sarcomas by genetics types (simple vs complex genomic profile) as part of the objective of identifying environmental risk factors.

Study design

The ETIOSARC study is a prospective multicenter population-based case-control study. This study is restricted to French geographical areas (further called districts) that meet at least one of these four criteria:

* Criteria 1: Districts covered by both a general cancer registry and a French Sarcoma Group (GSF-GETO) expert center from either the network of reference for soft-tissue sarcoma pathology (RRePS), the network of reference for bone sarcoma pathology (ResOs) or the clinical sarcoma network (NetSarc);
* Criteria 2: Districts including a coordinator center of any of the RRePS / NetSarc networks;
* Criteria 3: Districts covered by a general cancer registry that is expected to register more than 50 cases per year;
* Criteria 4: Districts adjacent to districts meeting criteria 1 and covered by a general cancer registry.

In total, 15 districts meet one of the four criteria, which represent approximatively 24% of the French population (2015 estimations from the national institute of statistics and economic studies, Insee). Nine districts meet criteria 1 (Gironde, Hérault, Haute-Vienne, Loire Atlantique, Calvados, Nord, Bas-Rhin and Doubs, Poitou-Charentes), two districts meet criteria 2 (Rhône and Val-de-Marne); two districts meet criteria 3 (Isère and Haut-Rhin) et two districts meet criteria 4 (Manche, Vendée).

Study population

Cases recruitment modalities

Patients will be recruited by specifically trained clinical research associate (CRA). In districts where a general cancer registry is active, the process of identifying incident sarcoma patients is well defined, which warrants the efficiency and exhaustiveness of the recruitment. However, poor survival for some cancer cases will not allow to rely on routine inclusion procedure and the registries will implement a rapid case ascertainment procedure to minimize the delay between diagnosis and enrollment and interview. Cases will be identified from pathology laboratories and multidisciplinary sarcoma tumor board (including sarcoma, gynecological, digestive, skin and bone tumor board). CRA will regularly contact laboratories and hospitals (within a three months window) to identify newly diagnosed sarcoma cases and to collect associated reports. The CRA will retrieve the clinical file in order to check inclusion and non inclusion criteria and to collect names and addresses of eligible patients and their physicians. Then, the CRA will contact the case's physicians in order to gather their clinical advice to include their patients in the study. In case of agreement, the CRA will contact the patients and ask them to participate. In case of oral agreement, he/she will arrange an interview to collect written consent and administer detailed questionnaire.

In Rhône and Val de Marne where no general cancer registry exists, the process of identifying incident sarcoma patients will largely rely on the existence of a RRePS/ResOS/NetSarc coordination center to facilitate the identification of new cases.

Regardless of the district, the diagnosis of all included cases will be systematically ascertained by an expert pathologist within the RRePS and ResOs networks following a standard procedure.

On a regular basis (at least once a month), the list of incident cases included in the RRePS/ResOS/NetSarc networks will be extracted from the shared databases. The list of cases identified by registries will be merged with the list of cases included in the RRePS/ResOS/NetSarc networks by the pathology sample reference number in order to collect diagnosis confirmation and to identify new but missed incident cases.

Controls selection

The selection of controls and the recruitment of cases will take place simultaneously. Every time a case will be diagnosed and identified, two controls will be randomly selected at that time from the electoral rolls of the same district as the case district of residence. For each case, a list of 20 potential controls with the same age (within a 5-year age group) and sex as the cases will be constituted in order to account for potential refusal. Calls to contact potential controls will be centralized and will be made by an investigator specifically trained to better understand the objectives of the study. First, this investigator will try to retrieve the phone number of the first potential control on the list and will contact him/her in order to gather his/her agreement to participate in this study. After five calls made at different schedules (e.g. in the evening on weekdays), if the potential control couldn't be reached, the investigator will send an information letter containing a reply coupon indicating phone number and schedule at which the person could be reach. If the reply coupon is not returned, or after 10 calls made at the phone number and the schedule indicated on the reply coupon, the first potential control will be considered as unreachable and then, the same procedure will be applied for the second potential controls on the list and so on until two controls per case agreed to participate to the study.

For each control agreeing to participate, an appointment will be made to collect written consent and to administer detailed questionnaire by a CRA.

All participants will give their informed written consent to participation, in line with French ethical guidelines.

Data collection

Data will be collected from self-questionnaire supplemented by a specific questionnaire. The self-questionnaire will permit to gather the complete occupational history (for each job held for at least 6 months) and residential history (for each place occupied for at least 6 months). During a face-to-face interview, the trained interviewer will check (complete if necessary) and supplement the self-administered questionnaire by a specific questionnaire with questions about demographic and socioeconomic characteristics, occupations of spouse and parents, leisure-time activities, reproduction, medical history, family history of cancer, diet, lifestyle factors such as tobacco smoking and alcohol consumption. The specific questionnaire will also collect additional occupational and residential information such as work tasks, work places, materials handled for each job held for at least 6 months and description of the environment of each residence places.

At the end of the interview, subjects (both cases and controls) will be invited to provide a saliva sample in order to obtain germline DNA.

In case of refusal to participate and if the subject agreed, data on demographic and socioeconomic characteristics will be collected in order to assess the potential selection bias that might occur due to the specific profile of non-respondent subjects.

Biological sampling and storage

Each participant will be asked to provide a salivary sample in order to obtain germline DNA. Salivary samples will be collected by the subjects themselves under instructions from the CRA, using DNA Genotek Oragene 575 collection kit. After collection, samples will be sent at the Biological Resources Center of the Bordeaux hospital university center "Bordeaux Biothèque Santé" for storage.

Determination of the sample size

Since our definition of environmental exposures is very broad, the sample size calculation has been based on various scenarios of exposure prevalence, from 5% (relevant for domestic, environmental but also some occupational exposures such as farmer in the general population) to 20% (relevant for some occupational exposures such as fibers). For a total sample size of 2000 cases and a 1:2 individually-matched design, considering a statistical power of 80% at a significance level of 5%, the minimum detectable odds ratio will be 1.39 and 1.21 under a exposure prevalence of 5% and 20%, respectively. Considering sub-types analyses, the four main histological types are GIST, liposarcoma, leiomyosarcoma and unclassified sarcoma, which account for 18%, 15%, 11% and 16% of sarcomas, respectively. Considering a sample size of 300 cases, the minimum detectable odds ratio will be 2.21 and 1.61 under an exposure prevalence of 5% and 20%, respectively. Typically in environmental epidemiology, the relative increases in disease risks due to environmental exposures are usually low around 1.5, thus, it is essential to recruit a minimum of 2000 cases in order to be able to perform sub-type analyses.

Statistical analysis

Relationship between case/control status and each exposure variable and 95% confidence intervals will be individually estimated using conditional logistic regression models. If necessary, a multilevel logistic model will be implemented in order to take into account the data variability due to the multicenter design and the various CRA that will administer the questionnaires.

Stratified histological sub-types analyses are also planned. Moreover, since sarcomas may be classified into four groups on a molecular basis (i.e. sarcomas with recurrent translocation, sarcomas with specific activating or inactivating mutations, sarcomas with MDM2 amplifications, and sarcomas with a complex genomic profile), the feasibility of classifying sarcomas by genetic types instead of by histological subtypes for the objective of identifying environmental risk factors will be explore. The underlying hypothesis is that the aetiology among these four molecular groups may be homogeneous.

Methods for coordinating the project and for quality control

This study is organized around three different centers or committees: a national coordination center, a steering committee, and local centers.

The national coordination center will be in charge of running routine operations, assisting participating local centers, guaranteeing the quality of the data collection, centralizing data, supervising the data coding and exposure assessment.

The steering committee's principal role will be to establish research priorities based on the availability of the data and the current scientific knowledge.

Local centers will be in charge of determining identification sources of cases in their districts and of collecting data. They will also transmit the collected data to the national coordination center.

Standardized procedures are written in a procedure manual to guarantee the quality of the collected data. Besides, a completion guide of the standardized questionnaire has been developed to assist CRA during interviews. A data manager will ensure that the study is conducted in compliance with the protocol. On a regular basis and as frequently as necessary, he/she will assess the quality of the collected data using several indicators: the average time spent by the CRA at the subject's home, the degree of completeness of the questionnaires by CRA, the ratio of included cases to expected cases, the average elapsed time between the identification of a case and the interview, the average elapsed time between case and control interviews, etc.

All collected data will be centralized in a single location, the University of Bordeaux (CREDIM, centre de Recherche et de Développement en Informatique Médicale).

ELIGIBILITY:
Inclusion Criteria:

* Cases

  * Patients diagnosed in the previous 6 months from identification with a primary and histologically confirmed malignant sarcoma including soft-tissue, visceral and bone sarcomas as defined by the WHO classification of bones and soft tissue sarcoma, fourth edition, 2013;
  * Diagnosed over a three-year period with an inclusion start date ranging from the 1st October 2018 to the 1st January 2020;
  * Living in the 15 districts participating to the study at the time of diagnosis
  * French nationality (due to control selection within electoral lists);
  * At least 18 years old at diagnosis;
  * Agreed to participate to the study with a signed informed consent;
* Controls

  * Subjects registered within the electoral rolls;
  * At least 18 years old at interview;
  * Living in the 15 districts participating to the study at the time of interview;
  * Agreed to participate to the study with a signed informed consent;

Exclusion Criteria:

* Cases

  * Patients with a known genetic predisposition to sarcoma such as Li-Fraumeni syndrome, Retinoblastoma syndrome, neurofibromatosis;
  * Kaposi's' sarcoma;
  * Protected adults' patients (aged of at least 18 years old) under guardianship by court order.
* Controls

  * Subject previously diagnosed with a primary and histologically confirmed malignant sarcoma including soft-tissue, visceral and bone sarcomas as defined by the WHO classification of bones and soft tissue sarcoma, fourth edition, 2013;
  * Protected adults' patients (aged of at least 18 years old) under guardianship by court order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases are defined as all incident patients with a diagnosis of primary sarcoma and histologically confirmed by an expert pathologist of the RRePS or ResOs networks in the 15 districts of France participating to this study.
  Two control subjects per case will be randomly selected from the French general population using electoral rolls and individually matched to case by age (by 5-year age group), sex and residential area.
Sampling Method: Probability Sample
Enrollment: 2237 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Odds ratios measuring the association between environmental exposures under study (environmental, occupational and lifestyle exposures) and sarcoma occurence | 1 year
  The relationship between case/control status and each exposure variable will be estimated by odds ratios and their 95% confidence intervals using conditional logistic regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Aude Lacourt, PhD, Principal Investigator — French National Institute of Health and Medical Research
Locations (10):
- France (10):
  - CHRU, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - CHU, Nantes
  - CHRU, Strasbourg
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data for both cases and controls will be made available under request to the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available at any time
Access Criteria: Data access requests will be reviewed by the steering committee Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Alexandrov LB, Stratton MR. Mutational signatures: the patterns of somatic mutations hidden in cancer genomes. Curr Opin Genet Dev. 2014 Feb;24(100):52-60. doi: 10.1016/j.gde.2013.11.014. Epub 2013 Dec 29. PMID 24657537
- [Background] Bisanti L, Maggini M, Raschetti R, Alegiani SS, Ippolito FM, Caffari B, Segnan N, Ponti A. Cancer mortality in ethylene oxide workers. Br J Ind Med. 1993 Apr;50(4):317-24. doi: 10.1136/oem.50.4.317. PMID 8494771
- [Background] Blair A, Zahm SH. Agricultural exposures and cancer. Environ Health Perspect. 1995 Nov;103 Suppl 8(Suppl 8):205-8. doi: 10.1289/ehp.95103s8205. PMID 8741784
- [Background] Briggs NC, Levine RS, Hall HI, Cosby O, Brann EA, Hennekens CH. Occupational risk factors for selected cancers among African American and White men in the United States. Am J Public Health. 2003 Oct;93(10):1748-52. doi: 10.2105/ajph.93.10.1748. PMID 14534232
- [Background] Burningham Z, Hashibe M, Spector L, Schiffman JD. The epidemiology of sarcoma. Clin Sarcoma Res. 2012 Oct 4;2(1):14. doi: 10.1186/2045-3329-2-14. PMID 23036164
- [Background] Downs TD, Crane MM, Kim KW. Mortality among workers at a butadiene facility. Am J Ind Med. 1987;12(3):311-29. doi: 10.1002/ajim.4700120307. PMID 3674024
- [Background] Ducimetiere F, Lurkin A, Ranchere-Vince D, Decouvelaere AV, Peoc'h M, Istier L, Chalabreysse P, Muller C, Alberti L, Bringuier PP, Scoazec JY, Schott AM, Bergeron C, Cellier D, Blay JY, Ray-Coquard I. Incidence of sarcoma histotypes and molecular subtypes in a prospective epidemiological study with central pathology review and molecular testing. PLoS One. 2011;6(8):e20294. doi: 10.1371/journal.pone.0020294. Epub 2011 Aug 3. PMID 21826194
- [Background] Ducimetiere F, Lurkin A, Ranchere-Vince D, Decouvelaere AV, Isaac S, Claret-Tournier C, Suignard Y, Salameire D, Cellier D, Alberti L, Bringuier PP, Blay JY, Ray-Coquard I. [Incidence rate, epidemiology of sarcoma and molecular biology. Preliminary results from EMS study in the Rhone-Alpes region]. Bull Cancer. 2010 Jun;97(6):629-41. doi: 10.1684/bdc.2010.1117. French. PMID 20504759
- [Background] Eriksson M, Hardell L, Adami HO. Exposure to dioxins as a risk factor for soft tissue sarcoma: a population-based case-control study. J Natl Cancer Inst. 1990 Mar 21;82(6):486-90. doi: 10.1093/jnci/82.6.486. PMID 2313720
- [Background] Grimalt JO, Sunyer J, Moreno V, Amaral OC, Sala M, Rosell A, Anto JM, Albaiges J. Risk excess of soft-tissue sarcoma and thyroid cancer in a community exposed to airborne organochlorinated compound mixtures with a high hexachlorobenzene content. Int J Cancer. 1994 Jan 15;56(2):200-3. doi: 10.1002/ijc.2910560209. PMID 8314301
- [Background] Guillou L, Aurias A. Soft tissue sarcomas with complex genomic profiles. Virchows Arch. 2010 Feb;456(2):201-17. doi: 10.1007/s00428-009-0853-4. PMID 20217954
- [Background] Hardell L, Eriksson M. The association between soft tissue sarcomas and exposure to phenoxyacetic acids. A new case-referent study. Cancer. 1988 Aug 1;62(3):652-6. doi: 10.1002/1097-0142(19880801)62:33.0.co;2-4. PMID 3390800
- [Background] Hoar SK, Blair A, Holmes FF, Boysen CD, Robel RJ, Hoover R, Fraumeni JF Jr. Agricultural herbicide use and risk of lymphoma and soft-tissue sarcoma. JAMA. 1986 Sep 5;256(9):1141-7. PMID 3801091
- [Background] Hoar Zahm S, Blair A, Holmes FF, Boysen CD, Robel RJ. A case-referent study of soft-tissue sarcoma and Hodgkin's disease. Farming and insecticide use. Scand J Work Environ Health. 1988 Aug;14(4):224-30. doi: 10.5271/sjweh.1928. PMID 3175554
- [Background] Hoppin JA, Tolbert PE, Flanders WD, Zhang RH, Daniels DS, Ragsdale BD, Brann EA. Occupational risk factors for sarcoma subtypes. Epidemiology. 1999 May;10(3):300-6. PMID 10230842
- [Background] Hossain A, McDuffie HH, Bickis MG, Pahwa P; Cross Canada Study of Pesticides and Health Researchers. Case-control study on occupational risk factors for soft-tissue sarcoma. J Occup Environ Med. 2007 Dec;49(12):1386-93. doi: 10.1097/JOM.0b013e318157d2f2. PMID 18231085
- [Background] Howe HL, Wingo PA, Thun MJ, Ries LA, Rosenberg HM, Feigal EG, Edwards BK. Annual report to the nation on the status of cancer (1973 through 1998), featuring cancers with recent increasing trends. J Natl Cancer Inst. 2001 Jun 6;93(11):824-42. doi: 10.1093/jnci/93.11.824. PMID 11390532
- [Background] IARC (2012). IARC Monographs on the Evaluation of Carcinogenic Risks to Humans, Vol. 100. A review of human carcinogens, part D: radiation. Lyon, IARC (International Agency for Research on Cancer)
- [Background] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. Chemical agents and related occupations. IARC Monogr Eval Carcinog Risks Hum. 2012;100(Pt F):9-562. No abstract available. PMID 23189753
- [Background] Karanian M, Coindre JM. [Fourth edition of WHO classification tumours of soft tissue]. Ann Pathol. 2015 Jan;35(1):71-85. doi: 10.1016/j.annpat.2014.11.003. Epub 2014 Dec 17. French. PMID 25532684
- [Background] Kogevinas M, Kauppinen T, Winkelmann R, Becher H, Bertazzi PA, Bueno-de-Mesquita HB, Coggon D, Green L, Johnson E, Littorin M, et al. Soft tissue sarcoma and non-Hodgkin's lymphoma in workers exposed to phenoxy herbicides, chlorophenols, and dioxins: two nested case-control studies. Epidemiology. 1995 Jul;6(4):396-402. PMID 7548348
- [Background] Landrigan PJ. Critical assessment of epidemiologic studies on the human carcinogenicity of 1,3-butadiene. Environ Health Perspect. 1990 Jun;86:143-7. doi: 10.1289/ehp.9086143. PMID 2205484
- [Background] Lurkin A, Ducimetiere F, Vince DR, Decouvelaere AV, Cellier D, Gilly FN, Salameire D, Biron P, de Laroche G, Blay JY, Ray-Coquard I. Epidemiological evaluation of concordance between initial diagnosis and central pathology review in a comprehensive and prospective series of sarcoma patients in the Rhone-Alpes region. BMC Cancer. 2010 Apr 19;10:150. doi: 10.1186/1471-2407-10-150. PMID 20403160
- [Background] Mathoulin-Pelissier S, Chevreau C, Bellera C, Bauvin E, Saves M, Grosclaude P, Albert S, Goddard J, Le Guellec S, Delannes M, Bui BN, Mendiboure J, Stoeckle E, Coindre JM, Kantor G, Kind M, Cowppli-Bony A, Hoppe S, Italiano A. Adherence to consensus-based diagnosis and treatment guidelines in adult soft-tissue sarcoma patients: a French prospective population-based study. Ann Oncol. 2014 Jan;25(1):225-31. doi: 10.1093/annonc/mdt407. Epub 2013 Nov 26. PMID 24285018
- [Background] Merletti F, Richiardi L, Bertoni F, Ahrens W, Buemi A, Costa-Santos C, Eriksson M, Guenel P, Kaerlev L, Jockel KH, Llopis-Gonzalez A, Merler E, Miranda A, Morales-Suarez-Varela MM, Olsson H, Fletcher T, Olsen J. Occupational factors and risk of adult bone sarcomas: a multicentric case-control study in Europe. Int J Cancer. 2006 Feb 1;118(3):721-7. doi: 10.1002/ijc.21388. PMID 16108052
- [Background] Pahwa P, McDuffie HH, Dosman JA, Robson D, McLaughlin JR, Spinelli JJ, Fincham S. Exposure to animals and selected risk factors among Canadian farm residents with Hodgkin's disease, multiple myeloma, or soft tissue sarcoma. J Occup Environ Med. 2003 Aug;45(8):857-68. doi: 10.1097/01.jom.0000083033.56116.c1. PMID 12915787
- [Background] Ray-Coquard I, Montesco MC, Coindre JM, Dei Tos AP, Lurkin A, Ranchere-Vince D, Vecchiato A, Decouvelaere AV, Mathoulin-Pelissier S, Albert S, Cousin P, Cellier D, Toffolatti L, Rossi CR, Blay JY. Sarcoma: concordance between initial diagnosis and centralized expert review in a population-based study within three European regions. Ann Oncol. 2012 Sep;23(9):2442-2449. doi: 10.1093/annonc/mdr610. Epub 2012 Feb 13. PMID 22331640
- [Background] Sathiakumar N, Delzell E, Austin H, Cole P. A follow-up study of agricultural chemical production workers. Am J Ind Med. 1992;21(3):321-30. doi: 10.1002/ajim.4700210305. PMID 1585943
- [Background] Savage SA, Mirabello L, Wang Z, Gastier-Foster JM, Gorlick R, Khanna C, Flanagan AM, Tirabosco R, Andrulis IL, Wunder JS, Gokgoz N, Patino-Garcia A, Sierrasesumaga L, Lecanda F, Kurucu N, Ilhan IE, Sari N, Serra M, Hattinger C, Picci P, Spector LG, Barkauskas DA, Marina N, de Toledo SR, Petrilli AS, Amary MF, Halai D, Thomas DM, Douglass C, Meltzer PS, Jacobs K, Chung CC, Berndt SI, Purdue MP, Caporaso NE, Tucker M, Rothman N, Landi MT, Silverman DT, Kraft P, Hunter DJ, Malats N, Kogevinas M, Wacholder S, Troisi R, Helman L, Fraumeni JF Jr, Yeager M, Hoover RN, Chanock SJ. Genome-wide association study identifies two susceptibility loci for osteosarcoma. Nat Genet. 2013 Jul;45(7):799-803. doi: 10.1038/ng.2645. Epub 2013 Jun 2. PMID 23727862
- [Background] Smith JG, Christophers AJ. Phenoxy herbicides and chlorophenols: a case control study on soft tissue sarcoma and malignant lymphoma. Br J Cancer. 1992 Mar;65(3):442-8. doi: 10.1038/bjc.1992.90. PMID 1558802
- [Background] Toro JR, Travis LB, Wu HJ, Zhu K, Fletcher CD, Devesa SS. Incidence patterns of soft tissue sarcomas, regardless of primary site, in the surveillance, epidemiology and end results program, 1978-2001: An analysis of 26,758 cases. Int J Cancer. 2006 Dec 15;119(12):2922-30. doi: 10.1002/ijc.22239. PMID 17013893
- [Background] Wibmer C, Leithner A, Zielonke N, Sperl M, Windhager R. Increasing incidence rates of soft tissue sarcomas? A population-based epidemiologic study and literature review. Ann Oncol. 2010 May;21(5):1106-11. doi: 10.1093/annonc/mdp415. Epub 2009 Oct 25. PMID 19858086
- [Background] Wingren G, Fredrikson M, Brage HN, Nordenskjold B, Axelson O. Soft tissue sarcoma and occupational exposures. Cancer. 1990 Aug 15;66(4):806-11. doi: 10.1002/1097-0142(19900815)66:43.0.co;2-u. PMID 2386907
- [Background] Woods JS, Polissar L, Severson RK, Heuser LS, Kulander BG. Soft tissue sarcoma and non-Hodgkin's lymphoma in relation to phenoxyherbicide and chlorinated phenol exposure in western Washington. J Natl Cancer Inst. 1987 May;78(5):899-910. PMID 3471999
- [Derived] Lacourt A, Amadeo B, Gramond C, Marrer E, Plouvier S, Baldi I, Blay JY, Coindre JM, de Pinieux G, Gouin F, Italiano A, Le Cesne A, Le Loarer F, Monnereau A, Pellegrin I, Penel N, Ray-Coquard I, Toulmonde M, Ducimetiere F, Mathoulin-Pelissier S; Etiosarc study group. ETIOSARC study : environmental aetiology of sarcomas from a French prospective multicentric population-based case-control study-study protocol. BMJ Open. 2019 Jun 18;9(6):e030013. doi: 10.1136/bmjopen-2019-030013. PMID 31217320